CLINICAL TRIAL: NCT03723408
Title: A Prospective Observational Study of Air Burden in Intravenous Tubing: Factors That Increase Patient Risk
Brief Title: Factors Increasing Air Burden in Intravenous Tubing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClearLine MD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLMD_CT_001
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Air Embolism; Air Leakage; Air Burden
MeSH Terms: conditions — Embolism, Air

STUDY DESIGN:
Intervention Model Description: An observational prospective trial was conducted in operating room settings across multiple study sites. 120 surgical patients undergoing a variety of interventional and surgical procedures were selected, representing multiple patient populations, case types and anesthesia setups. The ClearLine IV, a device that detects and removes air from IV tubing, was inserted into the IV circuit. Clinicians followed standard protocols. Blood warmers were used at the practitioner's discretion. IV fluid was administered at a constant flow rate or through a bolus given over 30-60 seconds per standard of care. The volume and duration of fluid administration was recorded, along with the frequency, duration and amount of air captured by ClearLine IV.
Masking Description: Three sites - Loma Linda Medical Center, Johns Hopkins, Miami Nicklaus Children's
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm post-approval study (Other): Single Arm post-approval study.
  Interventions: Device: ClearLine IV (formerly, AirPurge)

INTERVENTIONS:
Device: ClearLine IV (formerly, AirPurge) — Patient safety device that automatically and continuously detects and actively removes air from IV lines - protecting patients from dangerous air burden, air embolism, air infusions.
  Other Names: AirPurge

SUMMARY:
There is widespread acceptance that air in intravenous (IV) fluid tubing (lines) can pose a significant risk to patients.1 A rigorous literature search regarding sources of this air identified only anecdotal and non-clinical work regarding the presence and sources of air in IV tubing. Most published case studies have focused on air entrainment from accidental or inadvertent sources - empty IV fluid bags, incomplete priming of the tubing prior to infusion, and air-detection device failures, as examples.

The sources (and volume) of air inside IV tubing during common surgical procedures or interventions have yet to be studied prospectively. Understanding the frequency and magnitude of the presence of unintended air in IV tubing is the first step in devising potential avoidance strategies for eliminating unintended air in IV tubing. This study was designed to identify both the sources and magnitude of air that occurs in IV tubing during routine surgical procedures.

DETAILED DESCRIPTION:
Methods:

An observational prospective trial was conducted in operating room settings across multiple study sites. 120 surgical patients undergoing a variety of interventional and surgical procedures were selected, representing multiple patient populations, case types and anesthesia setups. The ClearLine IV, a device that detects and removes air from IV tubing, was inserted into the IV circuit. Clinicians followed standard protocols. Blood warmers were used at the practitioner's discretion. IV fluid was administered at a constant flow rate or through a bolus given over 30-60 seconds per standard of care. The volume and duration of fluid administration was recorded, along with the frequency, duration and amount of air captured by ClearLine IV.

ELIGIBILITY:
Inclusion Criteria:

* Any age - both pediatric and adult
* Weight equal to or greater than 5kg
* Surgical procedures
* Cardiac catherization procedures
* Minimum two hours procedure time

Exclusion Criteria:

* Patient weight less than 5 kg
* Procedures not involving surgery or cardiac catherization
* Procedures less than two hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
The frequency of air removed from intravenous tubing by ClearLine IV | 1 year
  The ClearLine IV data monitor measures the frequency (# of air masses) of air removed from IV lines
The amount of air removed from intravenous tubing by ClearLine IV | 1 year
  The ClearLine IV data monitor measures the amount (mL) of air removed from IV lines

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tirotta, MD, Principal Investigator — Nicklaus Children's Hospital; Jonathan Ho, MD, Principal Investigator — Johns Hopkins University; Davinder Ramsingh, MD, Principal Investigator — Loma Linda Medical Center

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03723408/Prot_SAP_000.pdf